CLINICAL TRIAL: NCT05834283
Title: Comparative Effects of Aerobic and Core Stability Exercise Training Program on Pain, Sleep and Quality of Life in Women With Endometriosis.
Brief Title: Aerobic vs Core Stability Exercise Training Program in Women With Endometriosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0522
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2023-04-28 (Actual); Status verified 2023-04

CONDITIONS: Endometriosis
Keywords: endometriosis; Aerobic exercises,; core stability,; Quality of life
MeSH Terms: conditions — Endometriosis | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- aerobic exercises (Experimental): This group will be received aerobic exercises 3 sessions per week for 8 weeks. Warm up phase: in which each participant will walk at 80 m/min at 0.0% grade for 5 mint.
  Active phase: treadmill speed will be increased to 147 m/min and grade will be increased gradually untill reached 25% grade for 20 mint.
  Cool down phase: in which the treadmil speed and grade will be decreased to 2.0miles/h and 0.0% grade during a cool down period consisted of 5 mint.
  Interventions: Other: aerobic exercises
- core stability exercises (Experimental): This group will be received core stability exercises 3 sessions per week for 8 weeks.
  All participants in both groups will be evaluated before and after the treatment programs.
  Lie on your back and place your feet on a wall so that your knees and hips are bent at 90 degrees angles. Tighten your abdominal muscles.
  Raise your head and shoulders off the floor. Return to the start position and repeat.
  Interventions: Other: core stability exercises

INTERVENTIONS:
Other: aerobic exercises — This group will be received aerobic exercises 3 sessions per week for 8 weeks. Warm up phase: in which each participant will walk at 80 m/min at 0.0% grade for 5 mint.
  Active phase: treadmill speed will be increased to 147 m/min and grade will be increased gradually untill reached 25% grade for 20 mint.
  Cool down phase: in which the treadmil speed and grade will be decreased to 2.0miles/h and 0.0% grade during a cool down period consisted of 5 mint.
  Arms: aerobic exercises
Other: core stability exercises — This group will be received core stability exercises 3 sessions per week for 8 weeks.
  All participants in both groups will be evaluated before and after the treatment programs.
  Lie on your back and place your feet on a wall so that your knees and hips are bent at 90 degrees angles. Tighten your abdominal muscles.
  Raise your head and shoulders off the floor. Return to the start position and repeat.
  Arms: core stability exercises

SUMMARY:
To compare the effects of aerobic and core stability exercise training program on pain, sleep and quality of life in women with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 24-45

  * Diagnosed patients with endometriosis
  * Pain lasting more than 6 months
  * Chronic pelvic pain
  * Infertility
  * Patients with dysmenorrhea.

Exclusion Criteria:

* Patients with the tubo- ovarian abscess.

  * Concomitment use of hormonal drugs.
  * Any malignancy
  * Impaired sensation..
  * Patients with Gynecological hemorrhage

Ages: 24 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Endometriosis is condition that occurs only in females
Enrollment: 30 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-01-08 (Actual); Study Completion 2023-03-15 (Actual)

PRIMARY OUTCOMES:
Numeric pain rating scale for pain | 8 weeks
  Numerical pain rating scale are the simplest and most commonly used scales. A tool used to help person rate the intensity of pain. The patients pick (verbal version) or draws a circle around (written version) the number that best describes the pain dimensions, usually intensity. The numeric pain rating scale for pain is a straight line with one end meaning no pain and the other end meaning worst pain
Endometriosis health profile questionnaire (EHP 30) for quality of life. | 8 weeks
  Endometriosis health profile questionnaire (EHP 30) is to evaluate the suitably self- report health status. It involves 30 items to identify the health status of patients with endometriosis. A core questionnaire which consists of five scales (pain, control and powerlessness, emotional well-being support and self-image)
Pittsburgh sleep quality index (PSQI) for sleep. | 8 weeks
  Pitts burgh sleep quality index (PSQI) is a self- rated questionnaire which asses the sleep quality and disturbance over a one-month time interval. It differentiates poor from good sleep quality. The PSQI is intended to be a standardized sleep questionnaire for clinicians and researchers to use with ease and is used for multiple populations. Clinical studies have found the PSQI to be reliable and valid in assessment of sleep problems to some degree

CONTACTS AND LOCATIONS:
Overall Officials: Hafiza Neelam, PPDPT, Principal Investigator — Riphah International University, Senior lecturer
Locations (1):
- Family Health Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vigano P, Parazzini F, Somigliana E, Vercellini P. Endometriosis: epidemiology and aetiological factors. Best Pract Res Clin Obstet Gynaecol. 2004 Apr;18(2):177-200. doi: 10.1016/j.bpobgyn.2004.01.007. PMID 15157637
- [Background] Bourdel N, Alves J, Pickering G, Ramilo I, Roman H, Canis M. Systematic review of endometriosis pain assessment: how to choose a scale? Hum Reprod Update. 2015 Jan-Feb;21(1):136-52. doi: 10.1093/humupd/dmu046. Epub 2014 Sep 1. PMID 25180023
- [Background] Ferrero S, Alessandri F, Racca A, Leone Roberti Maggiore U. Treatment of pain associated with deep endometriosis: alternatives and evidence. Fertil Steril. 2015 Oct;104(4):771-792. doi: 10.1016/j.fertnstert.2015.08.031. Epub 2015 Sep 10. PMID 26363387
- [Background] Chauvet P, Auclair C, Mourgues C, Canis M, Gerbaud L, Bourdel N. Psychometric properties of the French version of the Endometriosis Health Profile-30, a health-related quality of life instrument. J Gynecol Obstet Hum Reprod. 2017 Mar;46(3):235-242. doi: 10.1016/j.jogoh.2017.02.004. Epub 2017 Feb 7. PMID 28403920
- [Background] Cheong Y, William Stones R. Chronic pelvic pain: aetiology and therapy. Best Pract Res Clin Obstet Gynaecol. 2006 Oct;20(5):695-711. doi: 10.1016/j.bpobgyn.2006.04.004. Epub 2006 Jun 9. PMID 16765092